CLINICAL TRIAL: NCT05371444
Title: Effects of Control of Joint Degrees of Freedom in the Early Rehabilitation Post-stroke for the Recovery of Normal Movement (Non-compensatory) of the Upper Limb
Brief Title: Control of Degrees of Freedom Post-stroke for the Recovery of the Upper Limb
Acronym: DoF_UL_S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Principal Investigator, Pablo Burgos, Principal Investigator, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: hcuch_038; 11181337 (Other Grant/Funding Number: Fondecyt ANID)
Record Dates: First submitted 2021-04-26; First posted 2022-05-12 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Stroke
Keywords: True recovery; Neurorehabilitation; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The outcomes assessors will not now the arm to which each participant corresponds
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controlled DoF (Experimental): The treatment that this gruop will receive consist in a training with the exoskeleton that will restrict the DoF of the arm and trunk
  Interventions: Behavioral: Training with restriction of the DoF
- Non controlled DoF (Active Comparator): The treatment that this gruop will receive consist in a training with out the exoskeleton and without restriction of the DoF
  Interventions: Behavioral: Training without restriction of the DoF

INTERVENTIONS:
Behavioral: Training with restriction of the DoF — The intervention is based in the training of a single DoF of the upper extremity with restriction of the rest DoF of the arm and trunk that aren't being trained being restrained by an exoskeleton
  Arms: Controlled DoF
Behavioral: Training without restriction of the DoF — The intrevention is based in the training of the upper extremity movements without the restriction of DoF
  Arms: Non controlled DoF

SUMMARY:
The study's methodology will be a single-blind, multicenter, parallel-group randomized controlled trial (RCT). The sample consists of stroke patients (supratentorial ischemic and hemorrhagic stroke of anterior territory) between 18 and 80 years of age, separated into 2 groups of 20 participants. The experimental group called "controlled DoF", the control group 1 called "non controlled DoF". The "controlled DoF" group will use an exoskeleton that will restrict the movement of the trunk and upper limb to release only the joint to work in the plane of interest. The "non-controlled DoF" group will receive the same therapy time as the previous group but without any restriction of joint movements. The training will be functional with multiarticular and combined planes tasks. All groups receive the conventional rehabilitation of the health center (ideally 45 minutes 1 per day). Using motion sensors, clinical scales, and electroencephalography (EEG), the data will be obtained pre-intervention, post-intervention, and in a follow-up at 3 and 6 months.

DETAILED DESCRIPTION:
This proposal seeks to demonstrate if the control of joint degrees of freedom (DoF) of the trunk and upper limb is determinant during the early rehabilitation phase post-stroke (here from day 1 to day 28 or first month) for the recovery of upper limb movements without compensations and the normal brain control (true recovery).

The study's methodology will be a single-blind, multicenter, parallel-group randomized controlled trial (RCT). The sample consists of stroke patients (supratentorial ischemic and hemorrhagic stroke of anterior territory) between 18 and 80 years of age, separated into 2 groups of 20 participants. The experimental group called "controlled DoF", the control group 1 called "non controlled DoF". The "controlled DoF" group will receive for the initial 2 weeks, 2 hours of therapy, 5 times a week (2 sessions of 1 hour per day, 5 days) and the next 2 weeks, 2 hours of therapy, 3 times a week(2 sessions of 1 hour of therapy, 3 days), using an exoskeleton that will restrict the movement of the trunk and upper limb to release only the joint to work in the plane of interest. The training will be selective in an articulation plane with the biofeedback of active movements (or active-assisted) employing a video game controlled by an external movement sensor installed in the segment of interest. The "non-controlled DoF" group will receive the same therapy time as the previous group but without any restriction of joint movements. The training will be functional with multiarticular and combined planes tasks. All groups receive the conventional rehabilitation of the health center (ideally 45 minutes 1 per day). Using motion sensors, clinical scales, and electroencephalography (EEG), the data will be obtained pre-intervention, post-intervention, and in a follow-up at 3 and 6 months.

The expected results would show more functional improvements with less compensatory kinematics for therapy that control DoF than for the therapy without control of the DoF or for conventional therapy in acute post-stroke patients. About this result, the EEG connectivity analysis would show a lower interhemispheric inhibition of the motor areas and a greater frontal-parietal flow during reaching and manipulation tasks in the group with DoF control.

ELIGIBILITY:
Inclusion Criteria:

* (1) Clinical diagnosis of supratentorial ischemic stroke.
* (2) Time of onset <72 hours.
* (3) With alterations of the active voluntary movement of UL.
* (4) At least 3/8 DoF of the UE with MRC force scale of 3 or less.

Exclusion Criteria:

* (1) Cognitive impairment that prevents signing informed consent, following instructions and understanding procedures. (MoCA ≥ 18).
* (2) Musculoskeletal pathologies that prevent activities without pain or with limited ranges for the scope.
* (3) Severe visual impairment that does not allow the activities associated with the task.
* (4) Cerebellar o brainstem stroke.
* (5) Previous stroke leaving upper limb impairment.
* (6) Bilateral sensorimotor alterations.
* (7) Do not present alterations in functional clinical tests.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Normal movements Outcome. Kinematics of grasping and reaching 1 | At week 1
  Joint angles of the upper extremity in a water glass test
Normal movements Outcome. Kinematics of grasping and reaching 2 | At week 5
  Joint angles of the upper extremity in a water glass test
Normal movements Outcome. Kinematics of grasping and reaching 3 | At week 12
  Joint angles of the upper extremity in a water glass test
Normal movements Outcome. Kinematics of grasping and reaching 4 | At week 24
  Joint angles of the upper extremity in a glass test
Functioning Outcome 1 | At week 1
  Scale scores of Fugl Meyer Upper Limb test
Functioning Outcome 2 | At week 5
  Scale scores of Fugl Meyer Upper Limb test
Functioning Outcome 3 | At week 12
  Scale scores of Fugl Meyer Upper Limb test
Functioning Outcome 4 | At week 24
  Scale scores of Fugl Meyer Upper Limb test
Functioning Outcome - function of the arm1 | At week 1
  Scale scores of ARAT (Action Research Arm Test)
Functioning Outcome - function of the arm 2 | At week 5
  Scale scores of ARAT (Action Research Arm Test)
Functioning Outcome - function of the arm 3 | At week 12
  Scale scores of ARAT (Action Research Arm Test)
Functioning Outcome - function of the arm 4 | At week 24
  Scale scores of ARAT (Action Research Arm Test)
Functioning Outcome - daily life activities 1 | At week 1
  Scale scores of Barthel Index (independence in daily life activities)
Functioning Outcome - daily life activities 2 | At week 5
  Scale scores of Barthel Index (independence in daily life activities)
Functioning Outcome - daily life activities 3 | At week 12
  Scale scores of Barthel Index (independence in daily life activities)
Functioning Outcome - daily life activities 4 | At week 24
  Scale scores of Barthel Index (independence in daily life activities)
Functioning Outcome - quality of life 1 | At week 1
  Scale scores of EQ-5D (quality of life test)
Functioning Outcome - quality of life 2 | At week 5
  Scale scores of EQ-5D (quality of life test)
Functioning Outcome - quality of life 3 | At week 12
  Scale scores of EQ-5D (quality of life test)
Functioning Outcome - quality of life 4 | At week 24
  Scale scores of EQ-5D (quality of life test)
Connectivity Outcome 1 | At week 1
  Interhermispheric coherence of beta bands in the EEG.
Connectivity Outcome 2 | At week 5
  Interhermispheric coherence of beta bands in the EEG.
Connectivity Outcome 3 | At week 12
  Interhermispheric coherence of beta bands in the EEG.
Connectivity Outcome 4 | At week 24
  Interhermispheric coherence of beta bands in the EEG.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Maldonado, Doctor, Study Chair — University of Chile
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR, Analytic Code

DOCUMENTS (1):
  • Informed Consent Form (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT05371444/ICF_000.pdf